CLINICAL TRIAL: NCT04366752
Title: Thrombo Embolic Events in Critical Care Patients With Covid-19 Serious Acute Pneumopathy
Acronym: THROMBOCOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0036
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Pneumonia; ARDS; Hemostasis; Coagulation
Keywords: COVID-19; pneumonia; ARDS; venous ultrasound; hemostasis; coagulation
MeSH Terms: conditions — COVID-19; Pneumonia; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for coagulation and hemostasis analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: venous ultrasound — Venous ultrasound will be performed on patients once a week, every week from the day of admission in ICU until the day of patient discharge
Other: blood sample — blood sample for coagulation and hemostasis analysis will be withdrawn from artery catheter from the day of admission in ICU until the day of patient discharge

SUMMARY:
The understanding of haemostasis and inflammation cross-talk has gained considerable knowledge during the past decade in the field of arterial and venous thrombosis. Complex and delicately balanced interaction between coagulation and inflammation involve all cellular and humoral components. Elements of the coagulation system such as activated thrombin, fibrinogen or factor Xa may increase inflammation by promoting the production of pro-inflammatory cytokines, chemokines, growth factors and adhesion molecules that lead to a procoagulant state amplifying the pathological process. Recent evidence supports inflammation as a common pathogenic contributor to both arterial and venous thrombosis, giving rise to the concept of inflammation-induced thrombosis.

Patients with infection of COVID-19 and severe pneumoniae seem to have higher risk of thromboembolism. Very few data are available regarding the biological disorders of coagulation in these patients. Th purpose of this project is to analyze hemostasis and coagulation of patients with infection of COVID-19 and severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in medical ICU with pneumonia due to COVID-19 infection

Exclusion Criteria:

* patients< 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient hospitalized in CHU Amiens medical ICU with pneumonia due to COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Variation of thrombin time (in secondes) in Covid-19 patients with pneumonia admitted in ICU. | up to 6 weeks
  The reference range for the thrombin time is usually less than 20 seconds (ie, 15-19 seconds)
Variation of factor V concentration (U/dL) in Covid-19 patients with pneumonia admitted in ICU. | up to 6 weeks
  Variation of factor V concentration (U/dL) in Covid-19 patients with pneumonia admitted in ICU.
Variation of factor II concentration (U/dL) in Covid-19 patients with pneumonia admitted in ICU. | up to 6 weeks
  Variation of factor II concentration (U/dL) in Covid-19 patients with pneumonia admitted in ICU.
Variation of concentration of fibrin and fibrinogen degradation products (≥ 10 µgm/mL) in Covid-19 patients with pneumonia admitted in ICU. | up to 6 weeks
  Variation of concentration of fibrin and fibrinogen degradation products (≥ 10 µgm/mL) in Covid-19 patients with pneumonia admitted in ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No